CLINICAL TRIAL: NCT03403868
Title: Right Ventricular Haemodynamic Evaluation and Response to Treatment
Acronym: Rightheart I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Giessen (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Jan Grimminger, Principle Investigator, University of Giessen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 108/15
Record Dates: First submitted 2018-01-05; First posted 2018-01-19 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conductance catheter (Other): Contractility-measurement with conductance catheter (pressure-volume-catheter)
  Interventions: Diagnostic Test: conductance catheter

INTERVENTIONS:
Diagnostic Test: conductance catheter — pressure volume loops are assessed via a special catheter (Conductance catheter)

SUMMARY:
Mono-center Study to evaluate different multimodal functional parameter of the right ventricle in PAH-patients

DETAILED DESCRIPTION:
Mono-center-study tu evaluate functional parameters in cardiac MRI, conductance catheter (pressure-volume-loops), echocardiography and right heart catheter in PAH patients and to compare different multimodal parameters

ELIGIBILITY:
Inclusion Criteria:

* PH Nizza group 1 and patients without pulmonary hypertension after having the right heart catheter on clinical grounds
* ability to sign informed consent
* male and female between 18 to 85 years
* haemodynamic criteria:

  * Pulmonary vascular resistance (PVR) > 240 dyn x sec x cm-5
  * Mean Pulmonary artery pressure (mPAP) ≥ 25 mmHg for PAH patients
* normal haemodynamic in controls
* therapy-naive or at least since two months stabil therapy with approved drugs for PAH (Sildenafil, Tadalafil, Macitentan, Ambrisentan, Bosentan, Iloprost, Treprostinil, Riociguat).

Exclusion Criteria:

* therapy with positive inotropic drugs (dobutamin etc.)
* missing informed consent
* pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01; Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparibility of Ees (endsystolic elastance, which describes the right ventricular contractility) derived from conductance catheter, cMRI (cardiac magnetic resonance tomography) and 4D echocardiography | 12 weeks
  right ventricular contractility can be obtained via different methods, our aim is to compare the different methods.
  Ees is the endsystolic elastance which describes the contractility of the right ventricle

SECONDARY OUTCOMES:
dp/dt max and min from Pressure-Wire vs. Conductance Katheter | 12 weeks
  delta pressure/delta time is an indirect parameter of right ventricular contractility, which is load dependent
Comparibility of volumetry assessed via magnetic resonance tomography (MRI) and 4D echocardiography (ECHO) | 12 weeks
  Volumes (end-diastolic and endystolic) are measured via MRI and ECHO and compared with each other
Comparibility of pressures measured via pressure wire and conductance catheter | 12 weeks
  pressurewire measurements (high fidelity catheter) and conductance catheter (pressure volume catheter) are compared with each other

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Giessen, Giessen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kremer N, Rako Z, Douschan P, Gall H, Ghofrani HA, Grimminger F, Guth S, Naeije R, Rieth A, Schulz R, Seeger W, Tedford RJ, Vadasz I, Vanderpool R, Wiedenroth CB, Richter MJ, Tello K. Unmasking right ventricular-arterial uncoupling during fluid challenge in pulmonary hypertension. J Heart Lung Transplant. 2022 Mar;41(3):345-355. doi: 10.1016/j.healun.2021.11.019. Epub 2021 Dec 5. PMID 34972609
- [Derived] Tello K, Wan J, Dalmer A, Vanderpool R, Ghofrani HA, Naeije R, Roller F, Mohajerani E, Seeger W, Herberg U, Sommer N, Gall H, Richter MJ. Validation of the Tricuspid Annular Plane Systolic Excursion/Systolic Pulmonary Artery Pressure Ratio for the Assessment of Right Ventricular-Arterial Coupling in Severe Pulmonary Hypertension. Circ Cardiovasc Imaging. 2019 Sep;12(9):e009047. doi: 10.1161/CIRCIMAGING.119.009047. Epub 2019 Sep 10. PMID 31500448
- [Derived] Tello K, Dalmer A, Vanderpool R, Ghofrani HA, Naeije R, Roller F, Seeger W, Wilhelm J, Gall H, Richter MJ. Cardiac Magnetic Resonance Imaging-Based Right Ventricular Strain Analysis for Assessment of Coupling and Diastolic Function in Pulmonary Hypertension. JACC Cardiovasc Imaging. 2019 Nov;12(11 Pt 1):2155-2164. doi: 10.1016/j.jcmg.2018.12.032. Epub 2019 Mar 13. PMID 30878422
- [Derived] Tello K, Dalmer A, Axmann J, Vanderpool R, Ghofrani HA, Naeije R, Roller F, Seeger W, Sommer N, Wilhelm J, Gall H, Richter MJ. Reserve of Right Ventricular-Arterial Coupling in the Setting of Chronic Overload. Circ Heart Fail. 2019 Jan;12(1):e005512. doi: 10.1161/CIRCHEARTFAILURE.118.005512. PMID 30616360